CLINICAL TRIAL: NCT02690792
Title: Role of Mitochondrial Dysfunction in Non-Alcoholic Fatty Liver Disease
Brief Title: Effect of Vitamin E on Non-Alcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeffrey Browning (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Jeffrey Browning, Associate Professor of Internal Medicine, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 102010-180; R01DK087977-01A1 (NIH)
Record Dates: First submitted 2014-03-17; First posted 2016-02-24 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Healthy; NAFLD (Non-Alcoholic Fatty Liver Disease); NASH (Non-Alcoholic Steatohepatitis)
Keywords: Healthy; NAFLD; NASH; Liver Metabolism; Vitamin E
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NAFLD/NASH - Placebo (Placebo Comparator): In NAFLD/NASH Group: Identically appearing Placebo capsules given as double-blinded, randomized intervention as a comparator to Vitamin E intervention.
  Dosage: Placebo capsules. Two capsules by mouth each morning and two capsules by mouth each evening for 4 months.
  Interventions: Other: NAFLD/NASH - Placebo
- NAFLD/NASH - Vitamin E (Active Comparator): In NAFLD/NASH Group: Vitamin E capsules given as double-blinded, randomized intervention as a comparator to Placebo capsules intervention.
  Dosage: Vitamin E 200 IU/capsule. Two capsules by mouth each morning and two capsules by mouth each evening for 4 months.
  Interventions: Dietary Supplement: NAFLD/NASH - Vitamin E

INTERVENTIONS:
Other: NAFLD/NASH - Placebo — Placebo capsules, 2 capsules by mouth each morning and 2 capsules by mouth each evening for 4 months.
  Arms: NAFLD/NASH - Placebo
Dietary Supplement: NAFLD/NASH - Vitamin E — Vitamin E 200 IU capsule, 2 capsules by mouth each morning and 2 capsules by mouth each evening for 4 months.
  Arms: NAFLD/NASH - Vitamin E

SUMMARY:
One-third of the US population has non-alcoholic fatty liver disease (NAFLD) due to obesity and ~8 million of these individuals have a progressive form of the disease, non-alcoholic steatohepatitis (NASH). Currently, there are no noninvasive ways to determine which individuals with NAFLD will develop NASH. This is of medical importance since NASH can be a prelude to the development of end-stage liver disease.

The study of NAFLD has been limited by several factors, including the difficulties associated with studying liver metabolism in vivo in humans. Our group has pioneered new methods that use nuclear magnetic resonance (NMR) to measure intermediary hepatic metabolism in humans with a goal of directly studying the pathophysiology of bland steatosis and NASH. In this study, these noninvasive methods will be used to characterize and compare the metabolic alterations that accompany bland steatosis and NASH and test the hypothesis that detects if hepatic mitochondrial metabolism contribute to both disorders. Such characterization is fundamental to establishing a rational approach to the prevention and treatment of NAFLD and may provide simple, non-invasive methods to differentiate benign and progressive forms of NAFLD.

This proposal will be addressed via separate isotopic studies occurring at different time points during a prolonged fast. In subjects with NAFLD, these studies will be carried out before and after treatment with Vitamin E or placebo.

Healthy subjects will participate in initial baseline studies only without Vitamin E or placebo intervention.

The study is designed to harness the physiologic changes that occur with short- and long-term fasting to provide a rapid and cost-effective method to accomplish the aims of the application.

DETAILED DESCRIPTION:
Study Procedures (Healthy and NAFLD/NASH Subjects) Screening (Week -2) Prior to initiation of the timeline, all potential study participants will be evaluated by a research nurse to obtain informed consent, a brief medical history, height, weight, body mass index, waist/hip circumference, vital signs, approximately 20mls. of blood for screening labs and urine for analysis. NAFLD/NASH subjects with no available liver serologies will have an additional 25 mls of blood drawn. This visit will take approximately 60 minutes and will include a screening questionnaire for family history of disease, activities of daily living (ADL), and alcohol consumption. Diabetic subjects will also withhold their oral diabetic agent prior to the fasting screening labwork.

Teaching Visit: (Week -2 or prior to week -1): A research nurse will give diabetic subjects a 30-minute refresher course on diabetes that will include the signs and symptoms of hyper and hypoglycemia. A teaching booklet will be given to each diabetic subject. Some type 2 diabetic (T2DM) patients only on oral medication do not regularly check their blood sugar. If the patient does not have a glucometer, we will provide a glucometer, supplies and instructions for use by our diabetic study volunteers during their study participation.

Prior to the initiation of standardized diet, subjects will maintain their normal dietary routine. For three to four days prior to the protocol procedures, subjects will be placed on a standardized diet provided by the CTRC metabolic kitchen. In addition, participants will refrain from physical exercise at least 3 days prior to the procedures. Also, T2DM participants will withhold their oral diabetic agents for 3-4 days prior to the protocol procedures.

Phenotyping (Week -1) Participants will be asked to write down food and beverage consumption for three days prior to this visit. This food log will be turned into the dietician at the Clinical Translational Research Center (CTRC) for calculation of proteins, carbohydrates and fats in order to calculate a tailored 3.5 day meal plan to be consumed just prior to the overnight Fast.

Participants will be asked not to eat or drink anything after midnight prior to this visit in preparation for the day's study procedures.

Diabetic participants will withhold their oral diabetic agents for 3 days prior to the Phenotyping visit and the day of the visit. During this time, they will be instructed to check their blood glucose 30 minutes prior to each meal and at bedtime daily and will notify the research nurse or study physician if their blood glucose level is below 70 mg/dl or above 250 mg/dl.

Participants will arrive at the Advanced Imaging Research Center (AIRC) at approximately 8:30 AM. During the morning, participants will have measurements of liver fat in the 3 Tesla (3T) Magnetic Resonance (MR) scanner and measurement of their respiratory quotient (RQ) using an indirect calorimeter. Immediately following the scan, two intravenous catheters will be placed in preparation for the insulin/clamp study: an antecubital vein catheter to infuse dextrose and insulin and a dorsal hand vein catheter for blood sampling. The hand will be kept in a hot box at 70 °C for arterialization of venous blood. Three 10 ml. blood draws will be obtained for the baseline glucose level measurement, insulin infusate preparation, and blood chemistry analysis. At approximately 11:30 A.M., a primed continuous infusion of regular human insulin will be started for the duration of 2 hours. A 20% dextrose infusion will be started after 4 minutes of insulin infusion and adjusted to maintain euglycemia. A small amount of blood (1 ml.) will be drawn every 5 minutes for 2 hours to monitor plasma glucose concentration. The total amount of blood required for the whole procedure is approximately 80 mls. A urine specimen will be collected for determination of urinary glucose losses in the post-absorptive state. Approximately 3 healthy volunteers will have an additional measurement of liver fat after the insulin clamp to determine if changes are evident from the test. The participant will then be given a meal and discharged from the AIRC. The duration of this visit is approximately 7 hours.

Overnight Fast (Week 0) Diabetic participants will withhold their oral diabetic agents for 4 days prior to the Overnight Fast visit and the day of the visit. During this time, they will be instructed to check their blood glucose 30 minutes prior to breakfast and at bedtime daily and will notify the research nurse or study physician if their blood glucose level is below 70 mg/dl or above 250 mg/dl.

Four days prior to metabolic studies, participants will begin a tailored diet provided by the CTRC metabolic kitchen. The day prior to fasting studies, all participants will have the final meal at noon and begin fasting.

The following day they will arrive at the Advanced Imaging Research Center for a liver Magnetic Resonance Spectroscopy (MRS). Deuterium oxide (a.k.a. heavy water), the first stable isotope, will be administered according to the participant's weight in three divided doses.

Participants will receive carbon-13 labeled [U-13C]propionate (three 400 mg doses given by mouth over 1 hour). During the study, subjects will also be given 0.5% heavy water ad libitum. Subjects will undergo measurement of their respiratory quotient (RQ) using an indirect calorimeter just prior to the infusion protocol. Subjects will then have an intravenous catheter placed and an infusion of the stable isotopes carbon-13 labeled [3,4-13C2]glucose, carbon-13 labeled [1,2-13C]acetoacetate and carbon-13 labeled [3,4-13C]3-hydroxybutyrate initiated over two hours. During this period, 5 ml. blood draws will occur every hour to determine plasma non-esterified fatty acids (NEFA), ketones, glucose, insulin, and glucagon levels. At two hrs after initiation of the infusion, a 50 ml. blood draw will be performed to obtain samples for spectroscopic determination of the rate of ketogenesis and citrate oxidation in the citric acid (TCA) cycle. At the completion of study procedures, the stable isotope infusion will be stopped and participants will be sent to the CTRC outpatient clinic for Dual Energy x-Ray Absorptiometry (DEXA) to determine estimated total body fat measurement. After the DEXA, healthy subjects will be discharged to home; NAFLD subjects will be admitted to CTRC for liver biopsy, if needed.

The conclusion of the metabolic studies in week 0 marks the end of the study for control subjects, while NAFLD subjects will be initiated on Vitamin E or placebo therapy at this time point. All subjects will be given a meal and evaluated for stability (vital signs within normal limits) prior to discharge to home. The total amount of blood collected for overnight fasting studies will be less than 325 mls.

Follow-Up Visits (Weeks 4, 8, 12) Subjects will visit with the research nurse and/or Dr. Browning to monitor compliance with the vitamin E/placebo regime. At each follow-up visit, subjects will have blood collected (approximately 10mls.) per Table 1. Additionally, each volunteer will have an MRS to measure liver triglyceride content.

Phenotype Visit (Week 16) This is a repeat of the phenotype visit at Week -1.

Overnight Fast (Week 17) This is a repeat of the overnight fast at Week 0. All procedures, including the isotope studies will be the same.

ELIGIBILITY:
Inclusion Criteria:

NAFLD/NASH SUBJECTS

* Male and Female, Age 18-65 years of all racial and ethnic origins
* Hepatic steatosis by radiologic study with or without liver enzyme elevation
* BMI < 35 kg/m2
* English or Spanish language
* Females of childbearing potential must be willing to practice an acceptable form of birth control throughout the protocol
* May also have Type 2 Diabetes (T2DM) with:

Hemoglobin A1C < 8.5 % of total Prior, current or no oral antidiabetic medication usage

CONTROL SUBJECTS:

* Age 18-65 years.
* BMI ≤ 35 kg/m2
* English or Spanish language
* Females of childbearing potential must be willing to practice an acceptable form of birth control throughout the protocol
* May also have T2DM with:

Hemoglobin A1C < 8.5 % of total Prior, current or no oral antidiabetic medication usage

Exclusion Criteria:

ALL SUBJECTS:

* Diabetes type 1
* Diabetes type 2 with:

Hemoglobin A1C < 8.5 % of total Current or prior insulin usage

* Medications or conditions that confound the diagnosis of NAFLD
* Excessive alcohol intake (>30 g/day in men and >20 g/day in women)
* Chronic liver disease other than NAFLD/NASH
* Glucocorticoids
* Medications or conditions that alter hepatic metabolism
* Autoimmune disorders
* Current or chronic infection
* Other endocrine disorders
* Recent weight loss (> 10 lbs. within the past 3 months)
* Prescription weight-loss medications
* Medical conditions likely to increase the risk of intervention Renal insufficiency (creatinine > 1.4 mg/dL) Baseline metabolic acidosis Congestive heart failure
* Conditions or behaviors likely to affect the conduct of the study Pregnancy and breastfeeding confirmed by urine pregnancy test prior to all imaging or invasive procedure such as the euglycemic clamp, stable isotope studies, as well as prior to initiation of Vitamin E.
* Concurrent participation in another research project
* Inability to accept treatment assignment
* Major psychiatric disorder or substance abuse

CONTROL SUBJECTS (in addition to the above):

* Liver disease Elevated liver function tests Hepatic steatosis
* Metabolic syndrome Hypertriglyceridemia (fasting plasma triglycerides > 150 mg/dL). Systolic blood pressure > 140 mmHg Diastolic blood pressure > 80 mmHg
* Exercise above activities of daily living

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in Measurement of percentage of Liver Fat by MRI | baseline, 4 weeks, 8 weeks, 12 weeks, and 16 weeks
  Measurement of percentage of Liver Fat by MRI at baseline, 4 weeks, 8 weeks, 12 weeks, and 16 weeks.
Change in Measurement of Insulin Sensitivity via Hyperinsulinemic glucose clamp | 4 months
  Measurement of insulin sensitivity by glucose disposal rate (mg/Kg/min) via hyperinsulinemic glucose clamp @ baseline and 16 weeks.
Change in Measurement of glucose metabolism turnover by non-radioactive isotopic infusion and recovery | 4 months
  Measurement of glucose metabolism turnover (ug/Kg/min) in the liver by non-radioactive isotopic infusion and recovery @ baseline and 16 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D Browning, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fu X, Fletcher JA, Deja S, Inigo-Vollmer M, Burgess SC, Browning JD. Persistent fasting lipogenesis links impaired ketogenesis with citrate synthesis in humans with nonalcoholic fatty liver. J Clin Invest. 2023 May 1;133(9):e167442. doi: 10.1172/JCI167442. PMID 36928190